CLINICAL TRIAL: NCT02855333
Title: The Merendino Procedure for Benign or Early Malignant Lesions of the Distal Esophagus/Gastroesophageal Junction is Feasible, Safe and Provides Good QoL
Brief Title: Feasibility, Safety and QoL After Merendino Procedure
Acronym: MER
Status: Completed | Type: Observational
Sponsor: Kantonsspital Liestal (Other)
Responsible Party: Sponsor
Other Study IDs: KLiestal
Record Dates: First submitted 2016-07-13; First posted 2016-08-04 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Benign or Early Malignant Lesion of the Distal Esophagus or Gastro-esophageal Junction Requiring Surgical Resection
Keywords: Merendino procedure; Feasibility, Safety and QoL of the Merendino procedure

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Merendino Group (MER): Patients who underwent merendino procedure for benign or early malignant lesions of the distal esophagus/gastroesophageal junction Perioperative data and EORTC and QLQ-C30 / QLQ-OES24 questionnaire
  Interventions: Other: EORTC and QLQ-C30 / QLQ-OES24 questionnaire
- Control Group (CON): Patients who underwent alternative surgery for benign or early malignant lesions of the distal esophagus/gastroesophageal junction Perioperative data and EORTC and QLQ-C30 / QLQ-OES24 questionnaire
  Interventions: Other: EORTC and QLQ-C30 / QLQ-OES24 questionnaire

INTERVENTIONS:
Other: EORTC and QLQ-C30 / QLQ-OES24 questionnaire — EORTC and QLQ-C30 / QLQ-OES24 questionnaire was sent to patients to asses QoL after MER or CON procedure

SUMMARY:
The purpose of this study is to analyse retrospectively the early postoperative and functional outcome of patients (pts) after Merendino procedure for benign or early malignant lesions of the distal part of the esophagus or the gastroesophageal junction.

DETAILED DESCRIPTION:
Between 2004 and 2013, 14 pts had transhiatal resection of median 8 (6-10) cm of distal esophagus including the gastroesophageal junction. Locoregional lymphadenectomy was performed in all patients with (suspected) early adenocarcinoma. In case of vagus nerve resection, pyloromyectomy and cholecystectomy were done. A pediculated isoperistaltic jejunal segment of 15-18 cm length was interponed between esophageal stump and remaining stomach by end-to-side anastomoses. At least one postoperative contrast examination of the anastomoses was done in all pts. Quality of life was assessed by using the EORTC QLQ-OES18 survey, recording patients' general activity and condition and specific gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* alive
* MER or CON procedure
* informed consent
* CON patients were matched according to diagnosis, Age and ASA score

Exclusion Criteria:

* withdrawal of informed consent
* legal incapacity
* limitations in mental state or medical condition precluding questioning (only QoL data)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent Merendino procedure between 08/2004 and 02/2013 at the Kantonal Hospital of Baselland, Liestal (Switzerland) were included into the Merendino (MER) group. Considering indication for surgery, age, ASA score, and co-morbidities, patients who underwent gastrectomy during the same period were matched for control (CON) group.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) | up to 10 years after surgery
  EORTC QLQ-C30 and QLQ-OES24 questionnaire (global health status item, functional and symptom scale items)

SECONDARY OUTCOMES:
Intraoperative complications | up to 1 day after surgery
  Blood loss (ml), requirement for blood transfusion (units), operation time (min)
Postoperative complications | up to 100 days after surgery
  Morbidity (re-intervention rate, re-operation rate), in-hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A Maurer, MD, PhD, Study Director — Hirslanden
Locations (1):
- Kantonsspital Baselland, Liestal, Liestal, Basel-Landschaft, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zapletal C, Lorenz D. Quality of life after surgical treatment of early Barrett's cancer: a prospective comparison of the Ivor-Lewis resection versus the modified Merendino resection. A statistical hint: reply. World J Surg. 2014 Nov;38(11):3034. doi: 10.1007/s00268-014-2723-8. No abstract available. PMID 25189438
- [Background] Gotzky K, Jahne J. [Quality of life after operation for early Barrett's cancer: a prospective comparison of Ivor Lewis resection versus modified Merendino resection]. Chirurg. 2014 Sep;85(9):822. doi: 10.1007/s00104-014-2856-1. No abstract available. German. PMID 25123190
- [Background] Mangano A, Lianos GD, Rausei S, Boni L, Dionigi G. Quality of life after surgical treatment of early Barrett's cancer: a prospective comparison of the Ivor-Lewis resection versus the modified Merendino resection. A statistical hint. World J Surg. 2014 Nov;38(11):3033. doi: 10.1007/s00268-014-2624-x. No abstract available. PMID 24791672
- [Background] Zapletal Ch, Heesen Ch, Origer J, Pauthner M, Pech O, Ell Ch, Lorenz D. Quality of life after surgical treatment of early Barrett's cancer: a prospective comparison of the Ivor-Lewis resection versus the modified Merendino resection. World J Surg. 2014 Jun;38(6):1444-52. doi: 10.1007/s00268-013-2410-1. PMID 24378548
- [Background] Holscher AH, Vallbohmer D, Gutschow C, Bollschweiler E. Reflux esophagitis, high-grade neoplasia, and early Barrett's carcinoma-what is the place of the Merendino procedure? Langenbecks Arch Surg. 2009 May;394(3):417-24. doi: 10.1007/s00423-008-0429-9. Epub 2008 Nov 7. PMID 18989696